CLINICAL TRIAL: NCT04260685
Title: Intraoperative Lidocaine Versus Esmolol Infusion for Optimizing Surgical Field Visibility During Lumbar Discectomy
Brief Title: Lidocaine Versus Esmolol for Optimizing Surgical Field Visibility
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Zagazig University (Other Government)
Responsible Party: Principal Investigator, olfat abd elmoniem ibrahem, principle investigator, Zagazig University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 5901
Record Dates: First submitted 2020-01-21; First posted 2020-02-07 (Actual); Last update posted 2020-07-02 (Actual); Status verified 2020-06

CONDITIONS: Lumbar Disc Herniation
Keywords: esmolol; lidocaine; surgical field
MeSH Terms: conditions — Intervertebral Disc Displacement | interventions — Lidocaine; esmolol

STUDY DESIGN:
Intervention Model Description: Group L (lidocaine group) (n=35): the Patient will receive IV bolus of 1.5mg/kg lidocaine 1% over ten minutes followed by continuous infusion of 1.5mg/kg/h and will be terminated 10 minutes before the end of surgery.
  Group E(esmolol group) (n=35): the Patient will receive IV bolus of esmolol 0.5 mg/kg over ten minutes followed by continuous infusion of 100-300 ug/kg/min and will be terminated 10 minutes before the end of surgery.
Who Masked: Care Provider, Outcomes Assessor
Masking Description: the outcome assessor the surgeon
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- lidocaine (Active Comparator): the Patient will receive IV bolus of 1.5mg/kg lidocaine 1% over ten minutes followed by continuous infusion of 1.5mg/kg/h
  Interventions: Drug: Lidocaine
- esmolol (Active Comparator): the Patient will receive IV bolus of esmolol 0.5 mg/kg over ten minutes followed by continuous infusion of 100-300 ug/kg/min
  Interventions: Drug: Esmolol

INTERVENTIONS:
Drug: Lidocaine — IV bolus of 1.5mg/kg lidocaine 1% followed by continuous infusion of 1.5mg/kg/h
  Other Names: lignocaine
  Arms: lidocaine
Drug: Esmolol — IV bolus of esmolol 0.5 mg/kg followed by continuous infusion of 100-300 ug/kg/min
  Other Names: Brevibloc
  Arms: esmolol

SUMMARY:
Intra-operative blood loss is an important attribution and predictor of the lumbar spine surgery and patient outcome. Stripping the muscle off bone makes more exposed bleeding spine surface is one of causes for blood loss during lumbar surgeries. The importance to decrease the bleeding is to improve the surgical field visibility which provides technical ease for surgeon and decreases the surgical time besides maintaining the hemodynamic stability. In past, there were many trials to minimize surgical blood loss by different drugs such as Na Nitroprusside, magnesium sulfate, volatile anesthetics and beta-adrenergic antagonist.

DETAILED DESCRIPTION:
Sample size:

Assuming mean and standard deviation of mean arterial pressure in lidocaine group versus esmolol group is 90±27.9 versus 73± 22.5 so the sample size will be 70 (35 in each group ) using Open Epi program with confidence level 95%, power of test 80% All patients will be hospitalized and visited a day before the surgery, full history with physical examination and routine investigation will be done, the nature and complications of the study will be explained in detail to the patient and informed written consent will be obtained from every participant.

All patients will be kept nil orally 6 hours before the operation. All surgeries will be done by the same surgeon to decrease observer's bias. The surgeon and the outcome assessor (anesthesiologist collect the data) will be blinded to study drugs.

Using computer generated randomization table, each group consists of 35 patients.

ELIGIBILITY:
Inclusion Criteria:

* American society of anesthesiologist( ASA): I& II Physical status:
* Body Mass Index( BMI)=(25-35 kg/m2).
* Type of operations: lumbar discectomy.
* Written informed consent from the patient.

Exclusion Criteria:

* Patient refusal.
* .Altered mental state
* . Patients on beta-blockers or with a known history of allergy to study drugs.
* Hepatic, renal, Cardiovascular and respiratory diseases.
* Diabetic patients.
* Patients receiving anticoagulants.
* Previous spine surgery

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2020-02-04 (Actual); Primary Completion 2020-06-15 (Actual); Study Completion 2020-06-30 (Actual)

PRIMARY OUTCOMES:
The quality of surgical field visibility | from the start of surgery till the end of surgery
  using the surgical field rating (SFR) scale of six points proposed by (Fromme et al 1986) :
  Grade 0: No bleeding - virtually bloodless field. Grade 1: Slight bleeding so no suctioning required. Grade 2: Slight bleeding so occasional suctioning required. Grade 3: Low bleeding- frequent suctioning required; bleeding threatens surgical field some seconds after suction is removed.
  Grade 4: Moderate bleeding- frequent suctioning required, bleeding threatens surgical field directly after suctioning.
  Grade 5: Sever bleeding so constant suctioning required; bleeding appears faster than can be removed by suction; surgical field severely threatened and surgery hardly possible.
Mean arterial blood pressure | from induction of anesthesia till the end of surgery
  automatically invasive measured every 3 minutes , recorded every 15 minutes till the end

SECONDARY OUTCOMES:
heart rate | 15 minutes after the start of hypotensive agent
  heart rate
simplified postoperative nausea and vomiting | for the first 24 hours postoperative
  Postoperative nausea and vomiting impact scale score
surgeon satisfaction | "at completion of operation, an average 2 hours "
  Surgeon's satisfaction score
  1. Bad satisfaction.
  2. moderate satisfaction.
  3. Good satisfaction.
  4. excellent satisfaction
The need for blood transfusion | "through study completion, an average of four months".
  The number of patients need for blood transfusion: Acute blood loss more than 1,500 ml or 30% of blood volume is in need of blood transfusion
the amount of blood loss | from the beginning of surgery till the end of surgery, an average two hours"
  Blood loss= Hb (gdL/1) X V (mL)/Hbm (g/dL); Intraoperative blood volume loss (V)=blood in the suction container with adjustment for the used irrigating saline and the blood soaked by gauze pieces [4×4 soaked gauze piece =15 ml blood, completely soaked abdominal towel =150 ml blood].Hb= Hb concentration of suction container and Hbm=patient's mean hemoglobin concentration at the start

CONTACTS AND LOCATIONS:
Overall Officials: Olfat Ibrahem Amin, M.D, Principal Investigator — Zagazig University
Locations (1):
- Faculty of Medicine, Zagazig, Elsharkia, Egypt

IPD SHARING:
Plan to Share IPD: No